CLINICAL TRIAL: NCT06672432
Title: Preventing Perinatal Depression Using an App-based Cognitive Behavioral Therapy Program
Brief Title: Preventing Perinatal Depression with an App-Based CBT Program
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jintang County Maternal and Child Health Hospital (Other)
Collaborators: Chengdu Women's and Children's Central Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 20240511-1; 2024673 (Other Grant/Funding Number: Chengdu Health Commission)
Record Dates: First submitted 2024-10-31; First posted 2024-11-04 (Actual); Last update posted 2024-11-04 (Actual); Status verified 2024-10

CONDITIONS: Perinatal Depression; Disease Prevention
Keywords: Perinatal depression; cognitive behavioral therapy; iCBT

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Biostatisticians will be blinded to the study groups, ensuring that all results are analyzed and interpreted without bias.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- CareMom group (Experimental): The intervention program, CareMom, is a structured, 8-week digital intervention delivered through a WeChat mini-program in Chinese, developed by Shanghai Thoven Technology Co. Ltd., China, under the guidance of psychologists and psychiatrists. CareMom is designed to support perinatal mental health by providing daily challenges, educational content, and interactive exercises that target cognitive restructuring, behavioral activation, and worry management, key therapeutic components for alleviating symptoms of depression and anxiety. Participants in the intervention group will also receive standard perinatal care throughout the study. This includes routine prenatal check-ups, postpartum nursing care, and scheduled postnatal visits, ensuring that all participants receive the essential healthcare services typically provided during the perinatal period.
  Interventions: Other: CareMom (a mobile app-based 8-wekk cognitive behavioral therapy program)
- Control group (Active Comparator): The control group in this study will participate in an attention-matched, 8-week online relaxation training program delivered through a mobile application. Participants in the control group will also continue to receive standard perinatal care. This standard care is not altered or influenced by participation in the study, ensuring that all participants receive the usual care necessary for perinatal health.
  Interventions: Other: Matched Attention Control (a mobile app-based 8-week online relaxation training program)

INTERVENTIONS:
Other: CareMom (a mobile app-based 8-wekk cognitive behavioral therapy program) — The intervention is divided into daily tasks spread across eight weeks, with each day involving a variety of interactive elements such as videos, text-based content, guided reflections, and mental health check-ins. If the user misses a daily challenge, she can complete that challenge in the later days. Each week has a distinct focus that progressively builds the user's skills and understanding in managing emotional health. Tasks are designed to be short yet impactful, aiming to enhance engagement and adherence.
  Arms: CareMom group
Other: Matched Attention Control (a mobile app-based 8-week online relaxation training program) — This program is designed to mirror the structure and engagement level of the intervention group, providing participants with a similar amount of interaction and daily activities. Each day, participants in the control group will complete 1-2 daily tasks focused on relaxation techniques, such as breathing exercises, mindfulness meditation, and guided imagery. Each task is brief, approximately 3 minutes in duration, making it easy for participants to incorporate into their daily routine.
  Arms: Control group

SUMMARY:
The goal of this clinical trial is to learn if CareMom, a mobile app-based cognitive behavioral therapy program works to prevent perinatal depression among Chinese mothers. The main questions the trial aims to answer are:

1. Does CareMom lower depression scores after an 8-week intervention?
2. Does CareMom lower depression scores at 6 weeks after childbirth?
3. How satisfied are participants with CareMom?
4. What unfavorable events, if any, are associated with the use of CareMom?

Researchers will compare CareMom to a matched attention control (a mobile app-based program that offers participants a similar level of interaction and daily activities) to see if CareMom works to prevent perinatal depression.

Participants will:

1. Engage in the CareMom program or a relaxation training program every day for 8 weeks
2. Complete a series of online questionnaire tests before and after the 8-week intervention.
3. Report any discomfort experienced throughout the study period.

DETAILED DESCRIPTION:
A two-arm parallel randomised controlled trial of 290 pregnant women will be conducted at Jintang County Maternity and Child Health Hospital of Chengdu, China. Eligible women who consent to participate in the trial will be recruited at 20-24 weeks of gestation, and randomly allocated to either the intervention group (participate in a mobile app-based 8-week cognitive behavioral therapy program, named CareMom) or the control group (participate in a mobile app-based, attention-matched, 8-week relaxation training program) using a computer-generated random number. The primary outcomes are the changes in Edinburgh Postnatal Depression Scale (EPDS), Patient Health Questionnaire-9 (PHQ-9) and 7-item Generalized Anxiety Disorder (GAD-7) scores from From enrollment to the end of intervention at 8 weeks.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-45 years
* at 20-24 weeks of gestation
* at risk of depression but not experiencing severe depressive symptoms at recruitment, as indicated by an Edinburgh Postnatal Depression Scale (EPDS) score of between 5 and 12
* own a smartphone
* are able to independently engage with the program

Exclusion Criteria:

* have serious medical conditions or pregnancy complications that may affect their psychological condition, as determined by their medical doctor
* have a prior diagnosis of any mental disorders
* are currently or were recently (within the past six months) receiving any kinds of psychological services or treatments
* have a history of self-harm or suicide
* have any suicidal thoughts in the past 12 months
* experienced fetal deaths in the past 18 months

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 290 (Estimated)
Dates: Start 2024-11 (Estimated); Primary Completion 2025-07 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Changes in depression score at 6 weeks postpartum | From enrollment to 6 weeks postpartum
  Changes in Edinburgh Postnatal Depression Scale (EPDS) score. EPDS consists of 10 items rated on a four-point scale from 0 to 3, with a maximum score of 30, where higher scores indicate more severe depressive symptoms. We will use the Chinese version of EPDS in this study.
Changes in depression score at 6 weeks postpartum | From enrollment to 6 weeks postpartum
  Changes in Patient Health Questionnaire-9 (PHQ-9) score.The total scores of PHQ-9 range from 0 to 27, with a score of 10 or greater being the most common cut-off for screening major depressive disorder. We will use the Chinese version of the PHQ-9 in this study.
Changes in anxiety score at 6 weeks postpartum | From enrollment to 6 weeks postpartum
  Changes in Generalized Anxiety Disorder 7-item (GAD-7) score. GAD-7 consists of seven items, each rated on a score from 0 to 3. The total score ranges from 0 to 21, with higher scores reflecting more severe anxiety symptoms. In our study, the Chinese version of GAD-7 is applied.

SECONDARY OUTCOMES:
Changes in depression score at post-intervention | From enrollment to the end of intervention at 8 weeks
  Changes in Edinburgh Postnatal Depression Scale (EPDS) score. EPDS consists of 10 items rated on a four-point scale from 0 to 3, with a maximum score of 30, where higher scores indicate more severe depressive symptoms. We will use the Chinese version of EPDS in this study.
Changes in depression score at post-intervention | From enrollment to the end of intervention at 8 weeks
  Changes in Patient Health Questionnaire-9 (PHQ-9) score.The total scores of PHQ-9 range from 0 to 27, with a score of 10 or greater being the most common cut-off for screening major depressive disorder. We will use the Chinese version of the PHQ-9 in this study.
Changes in anxiety score at post-intervention | From enrollment to the end of intervention at 8 weeks
  Changes in Generalized Anxiety Disorder 7-item (GAD-7) score. GAD-7 consists of seven items, each rated on a score from 0 to 3. The total score ranges from 0 to 21, with higher scores reflecting more severe anxiety symptoms. In our study, the Chinese version of GAD-7 is applied.
Comparisons of satisfaction level | From enrollment to the end of intervention at 8 weeks
  Comparisons of Client Satisfaction Questionnaire (CSQ-8) results between the two groups. CSQ-8 consists of 8 items, resulting in scores that range from 8 to 32, with each item evaluated on a Likert scale; higher scores reflect greater levels of satisfaction.
Comparisons of adverse events | From enrollment to the end of intervention at 8 weeks
  Comparisons of adverse events between the two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Jintang County Maternity and Child Health Hospital, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No
IPD may not be shared due to privacy concerns and the need to protect sensitive information. However, we are open to sharing IPD upon reasonable request, ensuring that appropriate safeguards are in place to maintain participant confidentiality and comply with relevant regulations.

REFERENCES:
- [Derived] Tang L, Qing H, Li H, Liu C, Wang H, Sun Y, Tan Q, Wu Y, Xiao Y, Lai J, Wang L, Zhong L, Huang F, Li C. Reducing the risk of perinatal depression using an app-based cognitive behavioral therapy program: protocol of a randomized controlled trial. Front Psychiatry. 2025 Apr 14;16:1544753. doi: 10.3389/fpsyt.2025.1544753. eCollection 2025. PMID 40297330